CLINICAL TRIAL: NCT03228745
Title: The Health Impact of Mindfulness Based Stress Reduction on Total Knee Arthroplasty: A Pilot Study
Brief Title: The Health Impact of Mindfulness Based Stress Reduction on Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Renée El-Gabalawy, Dr., Assistant Professor, Staff Psychologist, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H2017:299
Record Dates: First submitted 2017-07-10; First posted 2017-07-25 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Total Knee Arthroplasty
Keywords: mindfulness based stress reduction; total knee arthroplasty; pre-operative
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre-operative MBSR (Experimental): Pre-operative MBSR is a condition where individuals will receive a pre-operative 8-week community-based MBSR course, which includes group classes lasting 2.5 hours a week, 45-minutes of home practice 6 days per week, a 1-hour orientation session at the beginning, and a full-day silent retreat at the end. During the orientation, participants will complete the study measures for this study.
  Interventions: Behavioral: Pre-operative MBSR
- treatment-as-usual (TAU) (No Intervention): The individuals in the TAU group will receive their treatment as usual.

INTERVENTIONS:
Behavioral: Pre-operative MBSR — A MBSR program typically consists of 8 weekly 2.5 hour sessions, home practice (typically 45 minutes per day, 6 days per week), and one day retreat. During the program, participants engage in a number of mindfulness practices (e.g., body scan, mindful movement, meditation) and discussions of their experiences, with the aim enhancing awareness to moment-to-moment experiences in a non-judging and accepting manner.
  Other Names: mindfulness based stress reduction
  Arms: pre-operative MBSR

SUMMARY:
Despite surgical success of total knee arthroplasty (TKA), reports of dissatisfaction and poor outcomes including increased pain, reduced function for daily activities, and compromised psychological health are common. Interventions to improve TKA outcomes are primarily education-focused, however there is little support for efficacy. Evidence suggests that mindfulness based stress reduction (MBSR) is effective for improving both physical and mental health, which are factors implicated in negative post-operative TKA outcomes. The efficacy of this empirically supported intervention on TKA outcomes has not been assessed. The proposed pilot study will conduct a randomized controlled trial to evaluate the feasibility and efficacy of pre-surgical MBSR on post-surgical outcomes. Post-operative pain (severity and catastrophizing), functioning (interference and illness impact), quality of life, emotional distress (anxiety and depression) and sleep will be assessed in pre-surgical MBSR and compared to treatment as usual. This pilot will provide an opportunity for TKA patients to receive an intervention that may improve outcomes. Further, it will provide insight into the relationship between pre-surgical MBSR and post-operative TKA outcomes, which will assist in the development of MBSR adaptations to less time intensive, and potentially more accessible, future offerings.

DETAILED DESCRIPTION:
Forty-five participants on the waitlist for a TKA will be recruited from Concordia Hospital Hip and Knee Institute - a facility that performs 800 TKA's per year. Participants will be divided into two groups: the pre-operative MBSR group (30 participants, divided into two MBSR groups), and the treatment-as-usual (TAU;15 participants). The individuals in the pre-operative MBSR group will receive a pre-operative 8-week community-based MBSR course taught by a certified instructor, which includes group classes lasting 2.5 hours a week, 45-minutes of home practice 6 days per week, a 1-hour orientation session at the beginning, and a full-day silent retreat at the end. During the orientation, participants will complete the study measures for this study. Two weeks prior to the surgery at the pre-anesthesia clinic, all patients will receive another set of short self-reported questionnaires. All patients will subsequently receive post-operative questionnaires at the following regularly scheduled post-operative appointments: 6-8 weeks after surgery, and at 6 month and 1 year follow-ups. Clinic personnel, who are blinded to assignment, will administer these measures with all other regularly distributed clinical measures. Clinic personnel will also review the chart to inform researchers as to what physical condition contributed to the need for a TKA. The TAU group will have the opportunity to enroll in an MBSR course following the completion of the study (after approximately 1 year), at no cost.

ELIGIBILITY:
Inclusion Criteria:

* on waitlist for first TKA

Exclusion Criteria:

* on waitlist for revision TKA
* taken a mindfulness course in the past 2 years
* not able to read or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Number of participants undergoing total knee arthroplasty who complete the mindfulness course MBSR to determine feasibility of this intervention | Up to 18 months
  Feasibility of MBSR intervention for TKA patients by determining the proportion of individuals who consent, are recruited, and complete the study.

SECONDARY OUTCOMES:
Cognitive function Patient- Reported Outcomes Measurements Information System (PROMIS) scales | Change in score from two weeks prior to surgery, week 6-8 post op, 6 month post-op, and 1 year post-op. If in the pre-operative MBSR group, also will complete these measures at the orientation of the MBSR program
  Brief self-report questionnaire with questions surrounding cognitive function
Fatigue PROMIS scale | Change in score from two weeks prior to surgery, week 6-8 post op, 6 month post-op, and 1 year post-op. If in the pre-operative MBSR group, also will complete these measures at the orientation of the MBSR program
  Brief self-report questionnaire with questions surrounding fatigue
Pain interference PROMIS scale | Change in score from two weeks prior to surgery, week 6-8 post op, 6 month post-op, and 1 year post-op. If in the pre-operative MBSR group, also will complete these measures at the orientation of the MBSR program
  Brief self-report questionnaire with questions surrounding pain interference
Pain behaviour PROMIS scale | Change in score from two weeks prior to surgery, week 6-8 post op, 6 month post-op, and 1 year post-op. If in the pre-operative MBSR group, also will complete these measures at the orientation of the MBSR program
  Brief self-report questionnaire with questions surrounding pain behaviour
Sleep disturbance PROMIS scale | Change in score from two weeks prior to surgery, week 6-8 post op, 6 month post-op, and 1 year post-op. If in the pre-operative MBSR group, also will complete these measures at the orientation of the MBSR program
  Brief self-report questionnaire with questions surrounding sleep disturbance
Psychosocial Illness Impact PROMIS scale | Change in score from two weeks prior to surgery, week 6-8 post op, 6 month post-op, and 1 year post-op. If in the pre-operative MBSR group, also will complete these measures at the orientation of the MBSR program
  Brief self-report questionnaire with questions surrounding psychosocial illness impact
Global health PROMIS scale | Change in score from two weeks prior to surgery, week 6-8 post op, 6 month post-op, and 1 year post-op. If in the pre-operative MBSR group, also will complete these measures at the orientation of the MBSR program
  Brief self-report questionnaire with questions surrounding global health
Anxiety PROMIS scale | Change in score from two weeks prior to surgery, week 6-8 post op, 6 month post-op, and 1 year post-op. If in the pre-operative MBSR group, also will complete these measures at the orientation of the MBSR program
  Brief self-report questionnaire with questions surrounding anxiety
Depression PROMIS scale | Change in score from two weeks prior to surgery, week 6-8 post op, 6 month post-op, and 1 year post-op. If in the pre-operative MBSR group, also will complete these measures at the orientation of the MBSR program
  Brief self-report questionnaire with questions surrounding anxiety
Pain Catastrophizing scale | Change in score from two weeks prior to surgery, week 6-8 post op, 6 month post-op, and 1 year post-op. If in the pre-operative MBSR group, also will complete these measures at the orientation of the MBSR program
  Brief self-report questionnaire surrounding pain catastrophizing
The benefit from mindfulness intervention assessed by the Five Facet Mindfulness Questionnaire | Change in score from two weeks prior to surgery, week 6-8 post op, 6 month post-op, and 1 year post-op. If in the pre-operative MBSR group, also will complete these measures at the orientation of the MBSR program
  Use a brief self-report questionnaire to determine if the participant's level of mindfulness increased as a result of the study

CONTACTS AND LOCATIONS:
Overall Officials: Renee El-Gabalawy, PhD, Principal Investigator — University of Manitoba; Jennifer Kornelsen, PhD, Principal Investigator — University of Manitoba; Eric Bohm, MD, Study Director — University of Manitoba; Corey Mackenzie, PhD, Study Director — University of Manitoba; Heather Macdonald, MD, Study Director — University of Manitoba; Gordon Asmundson, PhD, Study Director — University of Regina
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT03228745/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT03228745/SAP_001.pdf
  • Informed Consent Form (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT03228745/ICF_002.pdf